CLINICAL TRIAL: NCT00492921
Title: High-Dose Cyclophosphamide in Treating Patients With Acute Graft-Versus-Host Disease That Did Not Respond to Steroid Therapy
Brief Title: High-Dose Cyclophosphamide for Steroid Refractory GVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: J06116; P01CA015396 (NIH); P30CA006973 (NIH); NA_00003256 (Other: JHMIRB)
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Graft Versus Host Disease
Keywords: graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide

ARMS (3):
- Cyclophosphamide 50 (Experimental): Treatment with cyclophosphamide 50 mg/kg/d x 1 days.
  Interventions: Drug: Cyclophosphamide
- Cyclophosphamide 100 (Experimental): Treatment with cyclophosphamide 50 mg/kg/d x 2 days.
  Interventions: Drug: Cyclophosphamide
- Cyclophosphamide 150 (Experimental): Treatment with cyclophosphamide 50 mg/kg/d x 3 days.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide
  Other Names: Cy; CTX; Cytoxan

SUMMARY:
RATIONALE: High-dose cyclophosphamide may be an effective treatment for acute graft-versus-host disease that did not respond to steroid therapy.

PURPOSE: This phase II trial is studying the side effects, best dose, and how well high-dose cyclophosphamide works in treating patients with acute graft-versus-host disease that did not respond to steroid therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of high-dose cyclophosphamide in patients with steroid refractory acute graft-versus-host disease (GVHD).
* Determine the efficacy of this regimen at 28 days post-treatment in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive high-dose cyclophosphamide once daily for 1-4 days beginning on day 1 and filgrastim (G-CSF) subcutaneously once daily beginning on day 10 and continuing until blood counts recover.

Cohorts of 3-6 patients receive escalating doses of high-dose cyclophosphamide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed weekly for 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute graft-versus-host disease (GVHD) ≥ clinical grade II, that is steroid refractory

  * Steroid refractory GVHD is defined as GVHD that has progressed (increasing in grading) despite 49 hours of treatment with methylprednisolone of ≥ 2.0 mg/kg OR GVHD that has failed to improve (no change in grading stage) despite 4 days of treatment with methylprednisolone of ≥ 2.0 mg/kg
* Prior allogeneic hematopoietic stem cell transplantation using either bone marrow, peripheral blood stem cells, or cord blood OR prior donor lymphocyte infusion required
* Evidence of myeloid engraftment
* No chronic GVHD

PATIENT CHARACTERISTICS:

* ECOG (Eastern Cooperative Oncology Group) performance status (PS) 0-2 OR Karnofsky PS 60-100%
* ANC (absolute neutrophil count) > 500/mm³
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Must be geographically accessible
* No allergy or intolerance to cyclophosphamide or mesna
* No HIV positivity
* No mechanical ventilation
* No active bleeding (excluding gastrointestinal bleeding) or history of hemorrhagic cystitis
* No other uncontrolled illness including, but not limited to, the following:

  * Ongoing or active infection
  * Medical condition precluding patient from stopping azoles (e.g., fluconazole, itraconazole, or voriconazole) or other adequate antifungal therapy during cyclophosphamide administration
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Psychiatric illness/social situations that would preclude compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Bolanos-Meade, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclophosphamide 50 mg/kg: Treatment with cyclophosphamide 50 mg/kg/d x 1 day.
- Cyclophosphamide 100 mg/kg: Treatment with cyclophosphamide 50 mg/kg/d x 2 days.
- Cyclophosphamide 150 mg/kg: Treatment with cyclophosphamide 50 mg/kg/d x 3 days.
Period: Overall Study
Arm/Group | Cyclophosphamide 50 mg/kg | Cyclophosphamide 100 mg/kg | Cyclophosphamide 150 mg/kg
Started | 5 | 4 | 3
Completed | 4 | 4 | 2
Not Completed | 1 | 0 | 1
Not completed — Death | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Study site prefers to describe the study population as one set due to very small sample sizes for each arm.
Groups:
- Cyclophosphamide: Treatment with cyclophosphamide 50 mg/kg/d x 2 days, then dose adjusted according to continuous reassessment model according to toxicities until MTD found.
Arm/Group | Cyclophosphamide
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 38 [12 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of High-dose Cyclophosphamide as Determined by Number of Participants Who Tolerated Each Dose of Cyclophosphamide
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide 50 mg/kg | Cyclophosphamide 100 mg/kg | Cyclophosphamide 150 mg/kg
Number analyzed (Participants) | 5 | 4 | 3
Participants | 4 | 4 | 2

2. Primary Outcome: GVHD Response Rate
Description: Percentage of patients whose GVHD (as defined by Przepiorka criteria) responded to cyclophosphamide (complete response). Acute GVHD is defined by the Przepiorka criteria, which stages the degree of organ involvement in the skin, liver, and gastrointestinal (GI) tract, based on severity, with Stage 1+ being least severe and stage 4+ being the most severe. Grading of acute GVHD is as follows: Grade I (skin involvement stages 1+ to 2+, with no liver or GI involvement), Grade II (skin involvement stages 1+ to 3+, liver 1+, GI tract 1+), Grade III (skin involvement stages 2+ to 3+, liver 1+, GI tract 2+ to 4+), Grade IV (skin involvement stages 4+, Liver 4+).
Time Frame: Day 28
Population: This analysis excludes the two participants who died early because their responses were not assessed prior to death.
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide 50 mg/kg | Cyclophosphamide 100 mg/kg | Cyclophosphamide 150 mg/kg
Number analyzed (Participants) | 4 | 4 | 2
Participants | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: every week through Day 30
Description: The following events only were collected per the protocol's definition of an adverse event: unexpected adverse events that were attributed to the study drug by the investigator.
Arm/Group | Cyclophosphamide 50 mg/kg | Cyclophosphamide 100 mg/kg | Cyclophosphamide 150 mg/kg
All-Cause Mortality (participants affected / at risk) | 3/5 | 3/4 | 3/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/4 | 3/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide 50 mg/kg (N=5) | Cyclophosphamide 100 mg/kg (N=4) | Cyclophosphamide 150 mg/kg (N=3)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pain - abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No